CLINICAL TRIAL: NCT07386496
Title: The Role of 18F-PSMA PET in Prostate Cancer Diagnosis in Equivocal MRI: a Multi-center Randomised Controlled Trial
Brief Title: The Role of 18F-PSMA PET in Prostate Cancer Diagnosis in Equivocal MRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRE-2025.094
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMBINED arm (Experimental): In the COMBINED arm, additional pelvis-only 18F-PSMA-1007 PET-CT is performed within 6 months from mpMRI and before biopsy. Nuclear Medicine specialist interpreting PET-CT is blinded to clinical or MRI information.
  Interventions: Procedure: MRI+PSMA-guided approach
- MRI arm (Active Comparator): In the MRI arm, MRI-guided biopsy plus more than 12-core systematic biopsy will be performed.
  Interventions: Procedure: MRI-guided approach

INTERVENTIONS:
Procedure: MRI+PSMA-guided approach — MRI+PSMA-guided approach prostate biopsy
  Arms: COMBINED arm
Procedure: MRI-guided approach — MRI-guided approach prostate biopsy
  Arms: MRI arm

SUMMARY:
This study is a multi-center RCT to compare the clinically significant prostate cancer (csPCa) detection and/or change in clinical management in MRI guided (MRI arm) biopsy and MRI+18F-PSMA guided (Combined arm) biopsies in men with equivocal MRI prostate scans. If additional clinical value is shown by adding 18F-PSMA PET to equivocal MRI, then this should be the new standard of care.

DETAILED DESCRIPTION:
The investigators propose to conduct a phase III multi-center randomised controlled trial to evaluate the detection of clinically significant prostate cancer (csPCa) by MRI-guided biopsy approach (MRI arm) versus MRI+PSMA approach (COMBINED arm). Clinically significant prostate cancer (csPCa) is defined as prostate cancer classified as ISUP (International Society of Urogenital Pathology) Grade group 2 or higher. Patients with clinical suspicion of prostate cancer on MRI with PI-RADS (Prostate Imaging-Reporting and Data System, version 2.1) score 2 with red flag (PSA density >0.2 OR Prostate health index, PHI>35), PI-RADS 3, or PI-RADS 4 (and PSAd <0.1 OR PHI<35) will be randomised in a 1:1 manner to MRI arm or COMBINED arm. The detection rates of csPCa will be compared between arms. The study hypothesis is that COMBINED arm is superior to MRI arm in detecting csPCa and changing clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years of age
* Serum Prostate-specific antigen (PSA) 4-15 ng/mL, repeated at least once
* Prostate mpMRI done within 6 months
* MRI prostate with PI-RADS (11) scores of:

  * PI-RADS score 2 with red flag (PSA density >0.2 OR Prostate health index, PHI>35),
  * PI-RADS 3, OR
  * PI-RADS 4 with lower csPCa risks (PSAd <0.1 OR PHI<35)
* Normal Digital rectal examination
* Patient agrees for targeted and systematic prostate biopsy

Exclusion Criteria:

* Prostate biopsy within past 5 years
* Past or current history of prostate cancer
* Contraindicated to undergo PSMA PET-CT scan
* Contraindicated to prostate biopsy: active urinary tract infection, fail insertion of transrectal ultrasound probe into rectum (abdominal perineal resection, anal stenosis), fail to be placed in lithotomy position, uncorrectable coagulopathy, antiplatelet or anticoagulant which cannot be stopped (keep aspirin before and after biopsy is permitted)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 250 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of men with clinically significant Prostate cancer (csPCa) | When histology results available, at an expected average of 30 days post-biopsy
  ISUP Grade 2 or above prostate cancer diagnosed on biopsy
Proportion of men with additional csPCa detected only in PET targets which will affect clinical management | When histology results available, at an expected average of 30 days post-biopsy
  Determined by an independent and blinded panel with 3 urologists, including:
  * a change of nerve-sparing approach if radical prostatectomy is considered,
  * consideration or extent of focal therapy (partial gland ablation) of the prostate

SECONDARY OUTCOMES:
Proportion of men with csPCa detected in targeted and systematic biopsy | When histology results available, at an expected average of 30 days post-biopsy
  ISUP Grade 2 or above prostate cancer diagnosed on biopsy
Proportion of men with diagnosis of clinically insignificant prostate cancer | When histology results available, at an expected average of 30 days post-biopsy
  ISUP grade group 1 Prostate cancer diagnosed on biopsy
Proportion of men in combined arm with negative PET who could avoid a biopsy | When PET results available, at an expected average of 7 days post-scan
Correlation Between PET SUVmax of Targeted Lesion and Histologically Confirmed Clinically Significant Prostate Cancer (csPCa) | When histology results available, at an expected average of 30 days post-biopsy
  This outcome will quantify the correlation between:
  1. SUVmax of the PET-identified target lesion Measurement Tool: PET/CT scanner Unit of Measure: SUVmax (unitless)
  2. Histopathologic confirmation of csPCa in the corresponding biopsy cores Measurement Tool: Histology assessment by certified pathologist Unit of Measure: Presence or absence of csPCa (ISUP Grade 2 or above prostate cancer)
Proportion of men with post-biopsy adverse events within 30 days after biopsy | 30 days post biopsy
  The severity of Adverse event is grade by Clavien-Dindo classification
Health-related Quality of life scores | Assessed at baseline and at 30 days after intervention
  Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire.
  This instrument includes:
  1. Five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each scored on a 5-level scale from 1 to 5, where:
     * 1 = no problems
     * 5 = extreme problems / unable to perform (Higher scores indicate worse health status.)
  2. A Visual Analogue Scale (EQ-VAS) ranging from 0 to 100, where:
     * 0 = worst imaginable health
     * 100 = best imaginable health (Higher scores indicate better overall health.)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu PK, Teoh JY, Chan SY, Chu PS, Man CW, Hou SM, Ng CF. Role of PSA density in diagnosis of prostate cancer in obese men. Int Urol Nephrol. 2014 Dec;46(12):2251-4. doi: 10.1007/s11255-014-0826-7. Epub 2014 Sep 9. PMID 25201460
- [Background] Chiu PK, Teoh JY, Lee WM, Yee CH, Chan ES, Hou SM, Ng CF. Extended use of Prostate Health Index and percentage of [-2]pro-prostate-specific antigen in Chinese men with prostate specific antigen 10-20 ng/mL and normal digital rectal examination. Investig Clin Urol. 2016 Sep;57(5):336-42. doi: 10.4111/icu.2016.57.5.336. Epub 2016 Aug 31. PMID 27617315
- [Background] Chiu PK, Roobol MJ, Teoh JY, Lee WM, Yip SY, Hou SM, Bangma CH, Ng CF. Prostate health index (PHI) and prostate-specific antigen (PSA) predictive models for prostate cancer in the Chinese population and the role of digital rectal examination-estimated prostate volume. Int Urol Nephrol. 2016 Oct;48(10):1631-7. doi: 10.1007/s11255-016-1350-8. Epub 2016 Jun 27. PMID 27349564
- [Background] Gudmundsson J, Sulem P, Gudbjartsson DF, Masson G, Agnarsson BA, Benediktsdottir KR, Sigurdsson A, Magnusson OT, Gudjonsson SA, Magnusdottir DN, Johannsdottir H, Helgadottir HT, Stacey SN, Jonasdottir A, Olafsdottir SB, Thorleifsson G, Jonasson JG, Tryggvadottir L, Navarrete S, Fuertes F, Helfand BT, Hu Q, Csiki IE, Mates IN, Jinga V, Aben KK, van Oort IM, Vermeulen SH, Donovan JL, Hamdy FC, Ng CF, Chiu PK, Lau KM, Ng MC, Gulcher JR, Kong A, Catalona WJ, Mayordomo JI, Einarsson GV, Barkardottir RB, Jonsson E, Mates D, Neal DE, Kiemeney LA, Thorsteinsdottir U, Rafnar T, Stefansson K. A study based on whole-genome sequencing yields a rare variant at 8q24 associated with prostate cancer. Nat Genet. 2012 Dec;44(12):1326-9. doi: 10.1038/ng.2437. Epub 2012 Oct 28. PMID 23104005
- [Background] Chiu PK, Leow JJ, Chiang CH, Mok A, Zhang K, Hsieh PF, Zhu Y, Lam W, Tsang WC, Fan YH, Lin TP, Chan TY, Leung CH, Teoh JY, Chu PS, Zhu G, Ye DW, Wu HC, Tan TW, Tsu JH, Ng CF, Chiong E, Huang CY. Prostate Health Index Density Outperforms Prostate-specific Antigen Density in the Diagnosis of Clinically Significant Prostate Cancer in Equivocal Magnetic Resonance Imaging of the Prostate: A Multicenter Evaluation. J Urol. 2023 Jul;210(1):88-98. doi: 10.1097/JU.0000000000003450. Epub 2023 Apr 10. PMID 37036248
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Epstein JI, Egevad L, Amin MB, Delahunt B, Srigley JR, Humphrey PA; Grading Committee. The 2014 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma: Definition of Grading Patterns and Proposal for a New Grading System. Am J Surg Pathol. 2016 Feb;40(2):244-52. doi: 10.1097/PAS.0000000000000530. PMID 26492179
- [Background] Luo L, Zheng A, Chang R, Li Y, Gao J, Wang Z, Duan X. Evaluating the value of 18F-PSMA-1007 PET/CT in the detection and identification of prostate cancer using histopathology as the standard. Cancer Imaging. 2023 Nov 3;23(1):108. doi: 10.1186/s40644-023-00627-x. PMID 37924154
- [Background] Hoffmann MA, Muller-Hubenthal J, Rosar F, Fischer N, von Eyben FE, Buchholz HG, Wieler HJ, Schreckenberger M. Primary Staging of Prostate Cancer Patients with [18F]PSMA-1007 PET/CT Compared with [68Ga]Ga-PSMA-11 PET/CT. J Clin Med. 2022 Aug 29;11(17):5064. doi: 10.3390/jcm11175064. PMID 36078994
- [Background] Prive BM, Israel B, Janssen MJR, van der Leest MMG, de Rooij M, van Ipenburg JA, Jonker M, Peters SMB, de Groot M, Zamecnik P, Hoepping A, Bomers JG, Gotthardt M, Sedelaar JPM, Barentsz JO, van Oort IM, Nagarajah J. Multiparametric MRI and 18F-PSMA-1007 PET/CT for the Detection of Clinically Significant Prostate Cancer. Radiology. 2024 May;311(2):e231879. doi: 10.1148/radiol.231879. PMID 38771185
- [Background] Margel D, Bernstine H, Groshar D, Ber Y, Nezrit O, Segal N, Yakimov M, Baniel J, Domachevsky L. Diagnostic Performance of 68Ga Prostate-specific Membrane Antigen PET/MRI Compared with Multiparametric MRI for Detecting Clinically Significant Prostate Cancer. Radiology. 2021 Nov;301(2):379-386. doi: 10.1148/radiol.2021204093. Epub 2021 Aug 31. PMID 34463555
- [Background] Buteau JP, Moon D, Fahey MT, Roberts MJ, Thompson J, Murphy DG, Papa N, Mitchell C, De Abreu Lourenco R, Dhillon HM, Kasivisvanathan V, Francis RJ, Stricker P, Agrawal S, O'Brien J, McVey A, Sharma G, Levy S, Ayati N, Nguyen A, Lee SF, Pattison DA, Sivaratnam D, Frydenberg M, Du Y, Titus J, Lee ST, Ischia J, Jack G, Hofman MS, Emmett L. Clinical Trial Protocol for PRIMARY2: A Multicentre, Phase 3, Randomised Controlled Trial Investigating the Additive Diagnostic Value of [68Ga]Ga-PSMA-11 Positron Emission Tomography/Computed Tomography in Men with Negative or Equivocal Multiparametric Magnetic Resonance Imaging for the Diagnosis of Clinically Significant Prostate Cancer. Eur Urol Oncol. 2024 Jun;7(3):544-552. doi: 10.1016/j.euo.2023.11.008. Epub 2023 Dec 6. PMID 38061976
- [Background] Emmett L, Buteau J, Papa N, Moon D, Thompson J, Roberts MJ, Rasiah K, Pattison DA, Yaxley J, Thomas P, Hutton AC, Agrawal S, Amin A, Blazevski A, Chalasani V, Ho B, Nguyen A, Liu V, Lee J, Sheehan-Dare G, Kooner R, Coughlin G, Chan L, Cusick T, Namdarian B, Kapoor J, Alghazo O, Woo HH, Lawrentschuk N, Murphy D, Hofman MS, Stricker P. The Additive Diagnostic Value of Prostate-specific Membrane Antigen Positron Emission Tomography Computed Tomography to Multiparametric Magnetic Resonance Imaging Triage in the Diagnosis of Prostate Cancer (PRIMARY): A Prospective Multicentre Study. Eur Urol. 2021 Dec;80(6):682-689. doi: 10.1016/j.eururo.2021.08.002. Epub 2021 Aug 28. PMID 34465492
- [Background] Jain H, Sood R, Faridi MS, Goel H, Sharma U. Role of 68Ga-PSMA-PET/CT for the detection of primary prostate cancer prior to biopsy: a prospective study. Cent European J Urol. 2021;74(3):315-320. doi: 10.5173/ceju.2021.0084.R3. Epub 2021 Jul 8. PMID 34729219
- [Background] Padhani AR, Barentsz J, Villeirs G, Rosenkrantz AB, Margolis DJ, Turkbey B, Thoeny HC, Cornud F, Haider MA, Macura KJ, Tempany CM, Verma S, Weinreb JC. PI-RADS Steering Committee: The PI-RADS Multiparametric MRI and MRI-directed Biopsy Pathway. Radiology. 2019 Aug;292(2):464-474. doi: 10.1148/radiol.2019182946. Epub 2019 Jun 11. PMID 31184561
- [Background] Drost FH, Osses DF, Nieboer D, Steyerberg EW, Bangma CH, Roobol MJ, Schoots IG. Prostate MRI, with or without MRI-targeted biopsy, and systematic biopsy for detecting prostate cancer. Cochrane Database Syst Rev. 2019 Apr 25;4(4):CD012663. doi: 10.1002/14651858.CD012663.pub2. PMID 31022301
- [Background] Alberts AR, Roobol MJ, Verbeek JFM, Schoots IG, Chiu PK, Osses DF, Tijsterman JD, Beerlage HP, Mannaerts CK, Schimmoller L, Albers P, Arsov C. Prediction of High-grade Prostate Cancer Following Multiparametric Magnetic Resonance Imaging: Improving the Rotterdam European Randomized Study of Screening for Prostate Cancer Risk Calculators. Eur Urol. 2019 Feb;75(2):310-318. doi: 10.1016/j.eururo.2018.07.031. Epub 2018 Aug 3. PMID 30082150
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Background] Hamoen EHJ, de Rooij M, Witjes JA, Barentsz JO, Rovers MM. Use of the Prostate Imaging Reporting and Data System (PI-RADS) for Prostate Cancer Detection with Multiparametric Magnetic Resonance Imaging: A Diagnostic Meta-analysis. Eur Urol. 2015 Jun;67(6):1112-1121. doi: 10.1016/j.eururo.2014.10.033. Epub 2014 Nov 6. PMID 25466942
- [Background] Chiu PK, Roobol MJ, Nieboer D, Teoh JY, Yuen SK, Hou SM, Yiu MK, Ng CF. Adaptation and external validation of the European randomised study of screening for prostate cancer risk calculator for the Chinese population. Prostate Cancer Prostatic Dis. 2017 Mar;20(1):99-104. doi: 10.1038/pcan.2016.57. Epub 2016 Nov 29. PMID 27897172
- [Background] Chiu PK, Ng CF, Semjonow A, Zhu Y, Vincendeau S, Houlgatte A, Lazzeri M, Guazzoni G, Stephan C, Haese A, Bruijne I, Teoh JY, Leung CH, Casale P, Chiang CH, Tan LG, Chiong E, Huang CY, Wu HC, Nieboer D, Ye DW, Bangma CH, Roobol MJ. A Multicentre Evaluation of the Role of the Prostate Health Index (PHI) in Regions with Differing Prevalence of Prostate Cancer: Adjustment of PHI Reference Ranges is Needed for European and Asian Settings. Eur Urol. 2019 Apr;75(4):558-561. doi: 10.1016/j.eururo.2018.10.047. Epub 2018 Nov 2. PMID 30396635
- [Background] Chiu PK, Alberts AR, Venderbos LDF, Bangma CH, Roobol MJ. Additional benefit of using a risk-based selection for prostate biopsy: an analysis of biopsy complications in the Rotterdam section of the European Randomized Study of Screening for Prostate Cancer. BJU Int. 2017 Sep;120(3):394-400. doi: 10.1111/bju.13913. Epub 2017 Jun 5. PMID 28498624
- [Background] Carter HB, Hamper UM, Sheth S, Sanders RC, Epstein JI, Walsh PC. Evaluation of transrectal ultrasound in the early detection of prostate cancer. J Urol. 1989 Oct;142(4):1008-10. doi: 10.1016/s0022-5347(17)38971-1. PMID 2677409
- [Background] Culp MB, Soerjomataram I, Efstathiou JA, Bray F, Jemal A. Recent Global Patterns in Prostate Cancer Incidence and Mortality Rates. Eur Urol. 2020 Jan;77(1):38-52. doi: 10.1016/j.eururo.2019.08.005. Epub 2019 Sep 5. PMID 31493960
- [Background] Wong HF, Yee CH, Teoh JY, Chan SY, Chiu PK, Cheung HY, Hou SS, Ng CF. Time trend and characteristics of prostate cancer diagnosed in Hong Kong (China) in the past two decades. Asian J Androl. 2019 Jan 1;21(1):104-106. doi: 10.4103/aja.aja_75_18. No abstract available. PMID 30178778
- [Background] Chan SY, Ng CF, Lee KW, Yee CH, Chiu PK, Teoh JY, Hou SS. Differences in cancer characteristics of Chinese patients with prostate cancer who present with different symptoms. Hong Kong Med J. 2017 Feb;23(1):6-12. doi: 10.12809/hkmj164875. Epub 2016 Dec 9. PMID 27932742
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- See also: Hong Kong Cancer Statistics. — https://www3.ha.org.hk/cancereg/pdf/factsheet/2021/prostate_.pdf